CLINICAL TRIAL: NCT01935882
Title: A Double Blind Randomized Controlled Trial to Assess the Efficacy and Safety of Low Dose Primaquine for Clearance of Gametocytes in Asymptomatic Individuals Infected With P. Falciparum in Burkina Faso
Brief Title: Low Dose Primaquine for Clearance of Gametocytes
Acronym: LOPRIM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Radboud University Medical Center (Other); Centre national de recherche et de formation sur le paludisme (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOPRIM-1
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Malaria; Asymptomatic Malaria; Plasmodium Falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Artemether-Lumefantrine (Active Comparator): Artemether-Lumefantrine combination
  Interventions: Drug: Artemether-lumefantrine combination
- Artemether-Lumefantrine-Primaquine 0.25 (Experimental): Artemether-Lumefantrine with a single dose of 0.25mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine with a single dose of 0.25mg/kg primaquine
- Artemether-Lumefantrine-Primaquine 0.4 (Experimental): Artemether-Lumefantrine with a single dose of 0.4mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine with a single dose of 0.4mg/kg primaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine combination
  Arms: Artemether-Lumefantrine
Drug: Artemether-Lumefantrine with a single dose of 0.25mg/kg primaquine
  Arms: Artemether-Lumefantrine-Primaquine 0.25
Drug: Artemether-Lumefantrine with a single dose of 0.4mg/kg primaquine
  Arms: Artemether-Lumefantrine-Primaquine 0.4

SUMMARY:
Primaquine (PQ) is currently the only available drug that can clear mature transmission stages of P. falciparum parasites. PQ was previously shown to clear gametocytes that persist after artemisinin-combination therapy. However, there are safety concerns about the use of PQ at the currently recommended dose of 0.75mg/kg in individuals who are glucose-6-phosphate dehydrogenase (G6PD) deficient. PQ causes transient but significant haemolysis in G6PD deficient individuals; this side-effect is dose dependent. There are indications that a lower dosing of PQ may effectively reduce gametocyte carriage but the lowest efficacious dose for gametocyte clearance is currently unknown. Recently, the World Health Organization changed their recommendation to a low dose of primaquine, 0.25mg/kg. However, there is no direct evidence on the extent to which (low dose) PQ prevents malaria transmission to mosquitoes and what the lowest efficacious dose is.

In the current study we aim to identify the lowest efficacious dose of PQ in individuals with normal G6PD function. Children with asymptomatic malaria and normal G6PD enzyme function will be randomized to treatment with artemether-lumefantrine alone or in combination with low doses of PQ. All enrolled individuals will receive a full three-day course of AL, and will be randomized to receive a dose of primaquine or placebo with their fifth dose of AL. Efficacy will be determined based on gametocyte carriage during follow-up, measured by molecular methods. For a subset of participants with patent gametocytes, primaquine effect on infectivity to mosquitoes will be assessed by membrane feeding assays

ELIGIBILITY:
Inclusion Criteria:

1. Age > 2 years and <15 years
2. Weight over 10kg
3. P. falciparum parasitaemia >1,000 parasites and <200,000 parasites/µl
4. P. falciparum gametocytes detected by microscopy
5. Normal G6PD enzyme function
6. Informed consent by legally acceptable representative

Exclusion Criteria:

1. Enrolled in another study
2. Fever or history of fever in the last 24 hours
3. Evidence of severe illness/ danger signs
4. Known allergy to study medications
5. Hb < 8g/dL
6. Started menstruation
7. Pregnancy or breastfeeding
8. Antimalarials taken within the last 2 days
9. Primaquine taken within the last 4 weeks
10. Blood transfusion within the last 90 days
11. Non-falciparum malaria co-infection

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Gametocyte carriage | 14 days during follow-up
  Gametocyte prevalence at enrolment and on days 2, 3, 7, 10, 14 during follow-up.
  The duration of gametocyte carriage in days will be estimated.

SECONDARY OUTCOMES:
Transmission to Anopheles gambiae mosquitoes | day -1, day 3, day 7
  Mosquito membrane feeding assays will be used to determine the proportion of infected mosquitoes and the oocyst burden in infected mosquitoes.
Haematological recovery | 14 days during follow-up
  Haemoglobin concentration will be determined at enrolment and on days 2, 3, 7, 10 and 14 during follow-up. Haemoglobin concentration will be presented as grams per decilitre and as concentration relative to enrolment value.
Primaquine and lumefantrine pharmacokinetics | 7 days during follow-up
  The pharmacokinetic sampling will measure primaquine, lumefantrine and metabolites. Sampling involves 7 venous blood samples during the first 72 hours after treatment and a single later time point at day 7 post initiation of treatment. Drug plasma levels will be related to treatment arm and to the participant's Cytochrome P450 2D6 metabolizer status. CYP2D6 is an enzyme involved in primaquine metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Tiono, PhD, MD, Principal Investigator — Centre national de recherche et de formation sur le paludisme
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso

REFERENCES:
- [Derived] Goncalves BP, Pett H, Tiono AB, Murry D, Sirima SB, Niemi M, Bousema T, Drakeley C, Ter Heine R. Age, Weight, and CYP2D6 Genotype Are Major Determinants of Primaquine Pharmacokinetics in African Children. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02590-16. doi: 10.1128/AAC.02590-16. Print 2017 May. PMID 28289025
- [Derived] Goncalves BP, Tiono AB, Ouedraogo A, Guelbeogo WM, Bradley J, Nebie I, Siaka D, Lanke K, Eziefula AC, Diarra A, Pett H, Bougouma EC, Sirima SB, Drakeley C, Bousema T. Single low dose primaquine to reduce gametocyte carriage and Plasmodium falciparum transmission after artemether-lumefantrine in children with asymptomatic infection: a randomised, double-blind, placebo-controlled trial. BMC Med. 2016 Mar 8;14:40. doi: 10.1186/s12916-016-0581-y. PMID 26952094